CLINICAL TRIAL: NCT05124054
Title: Turkish Version of the Quality of Recovery-15 (QoR-15) Questionnaire
Brief Title: The Validity and Reliability of the Turkish Version of the Quality of Recovery-15 (QoR-15) Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, EMİNE ASLANLAR, Assistant professor, Selcuk University
Other Study IDs: QoR-15
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: to Evaluate the Feasibility, Reliability, Validity, and Responsiveness of the QoR-15T

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative recovery is a complex process influenced by various factors such as patients, surgical methods and anesthetic properties. Such factors can be accompanied by many negative situations. Previous studies evaluating recovery following anesthesia primarily evaluated the incidence of morbidity, mortality, adverse anesthesia-related outcomes, and changes in vital signs (1-4). These parameters are important, but the quality of recovery of patients has been neglected in most studies. Therefore, various patient-reported outcome measurement scales and tools have been developed (1,3-8). One of these scales is Stark et al. It is the QoR-15 questionnaire developed by in 2013 (4). QoR-15 aims to assess the quality of early recovery and emotional health of patients after surgery (4,6). It is a 15-item questionnaire assessing the patient's emotional state, physical comfort, psychological support, physical independence and pain. This one-page QoR-15 questionnaire has been shown to be highly valid and reliable in patients who have undergone general surgery (4).

QoR-15 has been verified and translated into many languages such as Japanese, French, Portuguese, Chinese, Swedish (13-17). It was reported in a systemic review that all translated versions of the QoR-15 had sufficient validity and reliability to assess the quality of postoperative recovery (19). However, an official Turkish version of the QoR-15 has not yet been developed or approved.

The aim of this study was to develop the Turkish version of the QoR-15 (QoR-15T) and to evaluate its validity, reliability and responsiveness for Turkish-speaking patients receiving general and regional anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* native turkish speaker
* scheduled elective surgery

Exclusion Criteria:

* with cognitive impairment,
* American Society of Anesthesiologists (ASA) physical condition IV or higher,
* patients with psychiatric disorders,
* history of alcohol or any other substance abuse
* patients expected to need postoperative mechanical ventilation (eg, cardiovascular surgery requiring cardiopulmonary bypass, microvascular reconstruction surgery for oral and maxillofacial cancer, etc.)
* Patients who are thought to be unable to answer the questionnaire due to a change in mental status or the need for sedation during the postoperative evaluation,
* patients who develop major complications after surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 65 who will undergo elective surgery and who is native Turkish speaker
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2021-12-04 (Actual); Primary Completion 2022-07-21 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
to evaluate the feasibility, reliability, validity, and responsiveness of the QoR-15T after surgery. | 5 min
  The QoR-15, a measurement tool to evaluate postoperative recovery in patients, consists of 15 items including pain, nausea, vomiting, and self-care status [9]. For each item, the patient is asked to express their status scoring from 0 to 10; therefore, the total score ranges from 0 to 150 points, with higher scores indicating better postoperative recovery. QoR-15 has been verified and translated into many languages such as Japanese, French, Portuguese, Chinese, Swedish.
  All translated versions of the QoR-15 were reported in a systemic review to have sufficient validity and reliability to assess the quality of postoperative recovery.The aim of this study is to develop the Turkish version of the QoR-15 (QoR-15T) and evaluate its validity, reliability and responsiveness for Turkish speaking patients receiving general and regional anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Aslanlar E, Aslanlar DA, Doganay C, Onal O, Sargin M, Cicekci F, Kara F, Kara I. The validity and reliability of the Turkish version of the quality of recovery-15 (QoR-15) questionnaire. Medicine (Baltimore). 2024 Apr 19;103(16):e37867. doi: 10.1097/MD.0000000000037867. PMID 38640327